CLINICAL TRIAL: NCT04282122
Title: Establishment of a Prospective Evaluation of Daily Practice Including the Individual Radiosensitivity Test to the Decision of Daily Practice
Brief Title: Clinical Database of Safe Personalized Adjuvant Breast Radiotherapy Based on Individual Radiosensitivity
Acronym: SAHARA-01
Status: Recruiting | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: PROICM 2018-09 BSA
Record Dates: First submitted 2019-10-21; First posted 2020-02-24 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; oncology; database; radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiotherapy — curative-intent radiotherapy

SUMMARY:
Severe but also moderate toxicities after curative-intent radiotherapy (RT), such as a poor cosmetic outcome following breast cancer can have a negative impact on quality of life and a marked effect on subsequent psychological outcome. Nevertheless, current practice standards commonly prescribe radiation dose and volume without regard to individual radiosensitivity.

In that context, a normal tissue radiosensitivity test that includes a rapid (72 h) radiosensitivity assay based on flow cytometric assessment of radiation-induced CD8 T-lymphocyte apoptosis (RILA) and other significant clinical parameters (multifactorial nomogram) was developed.

Omission of radiotherapy has been suggested when luminal A tumor subtype is combined with clinical and pathologic factors defining a subgroup of patients with a low risk of ipsilateral breast recurrence. In this group, the benefits of radiotherapy are small [6].

Reduction of the breast irradiated volume is also a possibility that has been tested and published using IORT, brachytherapy or external beam radiotherapy.

Hypofractionation has been adapted to breast cancer radiotherapy. Overall, all recent clinical trials [13, 14] showed only few late effects when hypofractionation was delivered to the whole breast (WB). These results reinforce the need of patients' selection using the NovaGray Breast® test.

Our hypothesis is therefore that the different techniques (volume reduction or hypofractionation) as well as radiotherapy omission will significantly reduce grade ≥2 bf+ in a personalized approach (driven by a predictive assay of late effects) compared to WB hypofractionation in a selected population at low risk of breast recurrence.

We would like to establish a prospective evaluation of daily practice including the individual radiosensitivity test to the decision of daily practice

DETAILED DESCRIPTION:
Severe but also moderate toxicities after curative-intent radiotherapy (RT), such as a poor cosmetic outcome following breast cancer can have a negative impact on quality of life and a marked effect on subsequent psychological outcome. Nevertheless, current practice standards commonly prescribe radiation dose and volume without regard to individual radiosensitivity.

In that context, a normal tissue radiosensitivity test that includes a rapid (72 h) radiosensitivity assay based on flow cytometric assessment of radiation-induced CD8 T-lymphocyte apoptosis (RILA) and other significant clinical parameters (multifactorial nomogram) was developed. The NovaGray Breast® test combines both a biological analysis (radio-induced lymphocyte apoptosis) and a predictive analysis, including external parameters related to the patient and her treatment. A negative predictive value (>90%) was found in case of high RILA taken alone and a sensitivity of 80% to detect the toxicity with an initial AUC of 0.61. In addition, including significant clinical parameters, the AUC was increased to 0.69. Moreover, a prognosis model with RILA alone to predict the probability to develop a toxicity and performance of the model was increased with the inclusion of significant clinical parameters (C-Harell 0.61 >> 0.69).

The NovaGray Breast® test is now validated after two prospective trials, one French (PHRC) and one European (Requite FP7). RILA and other factors have been confirmed to be independent factors that increase significantly the appearance of severe breast fibrosis. All these data have been merged into a nomogram allowing a predictive tool for daily clinical practice and then to customize radiotherapy techniques and indications.

In the meantime, several treatment modifications have been suggested to reduce late effects after breast radiotherapy:

Omission of radiotherapy has been suggested when luminal A tumor subtype is combined with clinical and pathologic factors defining a subgroup of patients with a low risk of ipsilateral breast recurrence. In this group, the benefits of radiotherapy are small [6]. In addition, low risk of recurrence was confirmed in randomized trials in a highly selected population. However, omitting radiotherapy and using intrinsic subtyping and clinical factors is a substantial change in care and could be driven by the risk of toxicity.

Reduction of the breast irradiated volume is also a possibility that has been tested and published using IORT, brachytherapy or external beam radiotherapy. The first two techniques are reserved for trained and expert centres but showed encouraging results with low toxicity rates and recurrences. The recent experience of external partial breast irradiation (EPBI) with twice daily fractions regimen showed an increase risk of late side-effects leading to use hypofractionated EPBI (hEPBI) once daily, 5 days a week. This regimen could only be used in case of selecting patients with NovaGray Breast®test without individual risk of late effects.

Hypofractionation has been adapted to breast cancer radiotherapy. Overall, all recent clinical trials showed only few late effects when hypofractionation was delivered to the whole breast (WB). Nevertheless, It has been shown in the TRANS-FAST trial a significant decrease of grade ≥2 bf+ for increasing values of RILA in the same extent than observed with conventional fractional schedules. These results reinforce the need of patients' selection using the NovaGray Breast® test.

ELIGIBILITY:
Inclusion Criteria:

1. Compliant women ≥ 65 years old.
2. Conservative breast cancer surgery.
3. T1-T2; N sentinel negative/N0.
4. Luminal A tumors.
5. Tumor negative margins.
6. Indication of whole breast irradiation only.
7. Extension evaluation of disease will be proven negative (M0).
8. Must be geographically accessible for follow-up.
9. Written and dated informed consent.
10. Affiliated to the French social security system.

Exclusion Criteria:

1. Patients with distant metastases.
2. Indications of node irradiation.
3. Synchronous bilateral breast cancer.
4. Patients treated by radical mastectomy.
5. Patients with neoadjuvant therapy.
6. Patients with previous or concomitant other (not breast cancer) malignancy within the past 3 years EXCEPT adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix. Patients who have had a previous other malignancy must have been disease free for at least three years.
7. Patients with other unstable or untreated non-malignant systemic diseases (cardiovascular, renal, hepatic, lung embolism, etc.) which would prevent prolonged follow-up.
8. Patients treated with systemic investigational drugs within the past 30 days

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients treated with safe adjuvant therapy by personalized radiation based on individual radiosensitivity after resection of breast tumor
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Acute and late breast fibrosis rate | Until the study completion: 5 years
  Describe the acute and late breast fibrosis rate in daily practice according to the individual radiosensitivity, assessed by the NovaGray RILA Breast® test

SECONDARY OUTCOMES:
Quality of life according to the EORTC QLQ-C30 | Until the study completion: 5 years
  Evaluate the quality of life according to the EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Céline BOURGIER, MD, Study Chair — Institut Régional du Cancer de Montpellier (ICM)
Locations (1):
- Institut Régional du Cancer de Montpellier, Montpellier, Occ, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bourgier C, Castan F, Riou O, Nguyen TD, Peignaux K, Lemanski C, Lagrange JL, Kirova Y, Lartigau E, Belkacemi Y, Rivera S, Noel G, Clippe S, Mornex F, Hennequin C, Gourgou S, Brengues M, Fenoglietto P, Ozsahin EM, Azria D. Impact of adjuvant hormonotherapy on radiation-induced breast fibrosis according to the individual radiosensitivity: results of a multicenter prospective French trial. Oncotarget. 2018 Mar 2;9(21):15757-15765. doi: 10.18632/oncotarget.24606. eCollection 2018 Mar 20. PMID 29644007
- [Background] Ozsahin M, Crompton NE, Gourgou S, Kramar A, Li L, Shi Y, Sozzi WJ, Zouhair A, Mirimanoff RO, Azria D. CD4 and CD8 T-lymphocyte apoptosis can predict radiation-induced late toxicity: a prospective study in 399 patients. Clin Cancer Res. 2005 Oct 15;11(20):7426-33. doi: 10.1158/1078-0432.CCR-04-2634. PMID 16243816
- [Background] Azria D, Gourgou S, Sozzi WJ, Zouhair A, Mirimanoff RO, Kramar A, Lemanski C, Dubois JB, Romieu G, Pelegrin A, Ozsahin M. Concomitant use of tamoxifen with radiotherapy enhances subcutaneous breast fibrosis in hypersensitive patients. Br J Cancer. 2004 Oct 4;91(7):1251-60. doi: 10.1038/sj.bjc.6602146. PMID 15328527
- [Background] Xiao B, Chen L, Ke Y, Hang J, Cao L, Zhang R, Zhang W, Liao Y, Gao Y, Chen J, Li L, Hao W, Sun Z, Li L. Identification of methylation sites and signature genes with prognostic value for luminal breast cancer. BMC Cancer. 2018 Apr 11;18(1):405. doi: 10.1186/s12885-018-4314-9. PMID 29642861
- [Background] Vaidya JS, Wenz F, Bulsara M, Tobias JS, Joseph DJ, Keshtgar M, Flyger HL, Massarut S, Alvarado M, Saunders C, Eiermann W, Metaxas M, Sperk E, Sutterlin M, Brown D, Esserman L, Roncadin M, Thompson A, Dewar JA, Holtveg HM, Pigorsch S, Falzon M, Harris E, Matthews A, Brew-Graves C, Potyka I, Corica T, Williams NR, Baum M; TARGIT trialists' group. Risk-adapted targeted intraoperative radiotherapy versus whole-breast radiotherapy for breast cancer: 5-year results for local control and overall survival from the TARGIT-A randomised trial. Lancet. 2014 Feb 15;383(9917):603-13. doi: 10.1016/S0140-6736(13)61950-9. Epub 2013 Nov 11. PMID 24224997
- [Background] Strnad V, Ott OJ, Hildebrandt G, Kauer-Dorner D, Knauerhase H, Major T, Lyczek J, Guinot JL, Dunst J, Gutierrez Miguelez C, Slampa P, Allgauer M, Lossl K, Polat B, Kovacs G, Fischedick AR, Wendt TG, Fietkau R, Hindemith M, Resch A, Kulik A, Arribas L, Niehoff P, Guedea F, Schlamann A, Potter R, Gall C, Malzer M, Uter W, Polgar C; Groupe Europeen de Curietherapie of European Society for Radiotherapy and Oncology (GEC-ESTRO). 5-year results of accelerated partial breast irradiation using sole interstitial multicatheter brachytherapy versus whole-breast irradiation with boost after breast-conserving surgery for low-risk invasive and in-situ carcinoma of the female breast: a randomised, phase 3, non-inferiority trial. Lancet. 2016 Jan 16;387(10015):229-38. doi: 10.1016/S0140-6736(15)00471-7. Epub 2015 Oct 19. PMID 26494415
- [Background] Olivotto IA, Whelan TJ, Parpia S, Kim DH, Berrang T, Truong PT, Kong I, Cochrane B, Nichol A, Roy I, Germain I, Akra M, Reed M, Fyles A, Trotter T, Perera F, Beckham W, Levine MN, Julian JA. Interim cosmetic and toxicity results from RAPID: a randomized trial of accelerated partial breast irradiation using three-dimensional conformal external beam radiation therapy. J Clin Oncol. 2013 Nov 10;31(32):4038-45. doi: 10.1200/JCO.2013.50.5511. Epub 2013 Jul 8. PMID 23835717
- [Background] Kunkler IH, Williams LJ, Jack WJ, Cameron DA, Dixon JM; PRIME II investigators. Breast-conserving surgery with or without irradiation in women aged 65 years or older with early breast cancer (PRIME II): a randomised controlled trial. Lancet Oncol. 2015 Mar;16(3):266-73. doi: 10.1016/S1470-2045(14)71221-5. Epub 2015 Jan 28. PMID 25637340
- [Background] Haviland JS, Owen JR, Dewar JA, Agrawal RK, Barrett J, Barrett-Lee PJ, Dobbs HJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Simmons S, Sydenham MA, Venables K, Bliss JM, Yarnold JR; START Trialists' Group. The UK Standardisation of Breast Radiotherapy (START) trials of radiotherapy hypofractionation for treatment of early breast cancer: 10-year follow-up results of two randomised controlled trials. Lancet Oncol. 2013 Oct;14(11):1086-1094. doi: 10.1016/S1470-2045(13)70386-3. Epub 2013 Sep 19. PMID 24055415